CLINICAL TRIAL: NCT06224686
Title: The Effect and Mechanism of Motor Imagery Based on Action Observation Treatment on Dysphagia in Wallenberg Syndrome
Brief Title: The Motor Imagery Based on Action Observation Treatment on Dysphagia in Wallenberg Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Wang (Other)
Responsible Party: Sponsor-Investigator, Le Wang, Master, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-PT310-01
Record Dates: First submitted 2024-01-06; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Lateral Medullary Syndrome; Deglutition Disorders
MeSH Terms: conditions — Lateral Medullary Syndrome; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): conventional dysphagia treatment and motor imagery based on action observation treatment
  Interventions: Other: conventional dysphagia treatment; Other: motor imagery based on action observation treatment
- The control group (Active Comparator): conventional dysphagia treatment
  Interventions: Other: conventional dysphagia treatment

INTERVENTIONS:
Other: conventional dysphagia treatment — Conventional dysphagia treatment included oropharyngeal muscle movement training, orofacial alternating hot and cold stimulation, Masako swallowing training, Mendelsohn maneuver, therapeutic ingestion training, intermittent oral-esophageal tube feeding, and low-frequency electrical stimulation of swallowing neuromusculature, etc., 30 min each time, once a day for 14 consecutive days.
Other: motor imagery based on action observation treatment — First, the therapist explained the purpose and principle of the intervention method to the patient, keeping the surrounding environment quiet and comfortable to avoid the patient's mood fluctuations due to external interference. Then start the treatment, the video recorded in advance was given to the patient to watch, the playback device is a ipad. The content includes lip and tongue muscle relaxation exercises, healthy people eating, chewing, swallowing, drinking and other images. At the same time, the guidance was played, which was consistent with the content in the video. The video was played 3 times consecutively for 30 min each time, once a day for 14 days.
  Arms: The experimental group

SUMMARY:
The goal of this clinical trial is to learn about on dysphagia in wallenberg syndrome. The main questions it aims to answer are:

* the efficacy of motor imagery based on action observation treatment in the rehabilitation of patients with dysphagia in Wallenberg syndrome.
* apply functional near infrared spectroscopy to explore the mechanism of action of this therapy.

Participants received conventional dysphagia treatment and motor imagery based on action observation treatment once a day for 14 days. Researchers compared the control group to see the effect and mechanism of motor imagery based on action observation treatment.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about on dysphagia in wallenberg syndrome. The main questions it aims to answer are:

* the efficacy of motor imagery based on action observation treatment in the rehabilitation of patients with dysphagia in Wallenberg syndrome.
* apply functional near infrared spectroscopy to explore the mechanism of action of this therapy.

Both groups received conventional dysphagia treatment, and the experimental group underwent the addition of motor imagery based on action observation treatment to the control group once a day for 14 days. Overall swallowing function was assessed before treatment and after 14 days of intervention. Meanwhile, the functional near infrared spectroscopy was used to detect changes in cerebral hemodynamics during the execution of volitional swallowing task and swallowing motor imagery.

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 18-80 years and right-handed;
* first onset, vital signs stable and conscious;
* the dysphagia confirmed by videofluoroscopic swallowing study;
* no cognitive impairment, the mini-mental state examination score: >17 for those with an illiterate education, >20 for those with an elementary education, and >24 for those with a secondary education and above;
* good motor imagery ability with kinesthetic and visual imagery questionnaire-10 score ≥25;
* cranial integrity without craniotomy and/or craniectomy;
* patient and/or his/her relative agrees and signs written informed consent.

Exclusion Criteria:

* combined ischemic foci at other sites;
* presence of organic swallowing dysfunction or pre-existing dysphagia due to Parkinson's disease, dementia, and others;
* severe cardiac, pulmonary, hepatic, and renal insufficiency and vital organ failure;
* significant psychological disorders such as anxiety and depression;
* infected or broken skin on the head;
* poorly controlled epilepsy;
* poor patient compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
standardized swallowing assessment | day 1 and day 14
  The standardized swallowing assessment was used to assess the improvement of overall swallowing function, it has a maximum score of 46 and a minimum score of 18, with lower scores indicating better swallowing function.
cortical activation during volitional swallowing | day 1 and day 14
  The functional near infrared spectroscopy system (Nirsmart, Danyang Huichuang Medical Equipment Co., Ltd., China) was used to detect changes in cerebralhemodynamics during the execution of volitional swallowing task.
cortical activation during swallowing motor imagery | day 1
  The functional near infrared spectroscopy system (Nirsmart, Danyang Huichuang Medical Equipment Co., Ltd., China) was used to detect changes in cerebralhemodynamics during the whole swallowing motor imagery.

SECONDARY OUTCOMES:
Murray secretion scale | day 1 and day 14
  The severity of Murray secretion scale was measured using a grade of 0-3, patients without obvious saliva accumulation are scored as MSS grade 0, whereas patients who had secretions in the laryngeal vestibule at the start of the exam were assigned grade 3.
yale pharyngeal residue severity rating scale | day 1 and day 14
  Yale pharyngeal residue severity rating scale scores were measured using a 5-point ordinal scale: Ⅰ = none, Ⅱ = trace, Ⅲ = mild, Ⅳ = moderate, Ⅴ = severe.
Rosenbek penetration-aspiration scale | day 1 and day 14
  The highest PAS score is 8 and the lowest is 1 (1 = no entry of material into the airway; 2 - 5 = penetration of material past the laryngeal additus into the supraglottic space and traveling as far as the true vocal folds; 6 - 8 = tracheal aspiration of material below the true vocal folds).
swallowing-quality of life | day 1 and day 14
  Swallowing-quality of life has a score range of 44 - 220, with lower scores indicating poorer swallowing function and poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zeng, Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to the hospital's confidentiality regulations regarding trial data but are available from the corresponding author on reasonable request.